CLINICAL TRIAL: NCT07012590
Title: Morphine and Dexmedetomidine as Adjuvants to Bupivacaine in Ultrasound-guided Erector Spinae Plane Block for Open Subcostal Renal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ayman Essam Kaka, Resident of Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine, Kafr Elsheikh University, Kafr Elsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-525
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Morphine; Dexmedetomidine; Adjuvants; Bupivacaine; Ultrasound; Erector Spinae Plane Block; Open Subcostal Renal Surgeries
MeSH Terms: interventions — Morphine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morphine group (Experimental): Patients received erector spinae plane block with morphine 2 mg as an adjuvant to bupivacaine 30 ml 0.25%.
  Interventions: Drug: Morphine
- Dexmedetomidine group (Experimental): Patients received erector spinae plane block with dexmedetomidine 100 µg as an adjuvant to bupivacaine 30 ml 0.25%.
  Interventions: Drug: Dexmedetomidine
- Control group (Active Comparator): Patients received erector spinae plane block with bupivacaine 30 ml 0.25% only.
  Interventions: Other: Erector spinae plane block

INTERVENTIONS:
Drug: Morphine — Patients received erector spinae plane block with morphine 2 mg as an adjuvant to bupivacaine 30 ml 0.25%.
  Arms: Morphine group
Drug: Dexmedetomidine — Patients received erector spinae plane block with dexmedetomidine 100 µg as an adjuvant to bupivacaine 30 ml 0.25%.
  Arms: Dexmedetomidine group
Other: Erector spinae plane block — Patients received erector spinae plane block with bupivacaine 30 ml 0.25% only.
  Arms: Control group

SUMMARY:
This study aimed to compare the analgesic efficacy between morphine and dexmedetomidine as adjuvants to bupivacaine in ultrasound-guided erector spinae plane block for open subcostal renal surgeries.

DETAILED DESCRIPTION:
The postoperative pain that occurs because of the wide flank incision ranges from a moderate to severe intensity and, in some patients, can become chronic.

The erector spinae plane block (ESPB) is a novel interfascial plane technique, aiming to block the dorsal and ventral rami of the spinal nerves to provide visceral and somatic multi-dermatomal analgesia of the cervical, thoracic, and lumbar levels.

Adjuvants to local anesthetics, such as morphine and dexmedetomidine, can be used to improve the quality and duration of peripheral nerve block effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient's approval.
* Age: 20 - 65 years.
* Physical Status: American Society of Anesthesiologists (ASA) I & II.
* Patients undergoing open subcostal renal surgeries.

Exclusion Criteria:

* Patient refusal.
* Age: >65 and <20 years.
* Allergy to Dexmedetomidine, local anesthetics, systemic opioids, and any of the drugs included in the multimodal perioperative pain protocol.
* Patient with coagulation disorders.
* Chronic pain syndromes and patients with chronic opioid use are defined as use of regular daily doses of systemic narcotics for the past 6 months before the surgery.
* Body mass index of 35 kg/ m2 or more.
* Physical Status: American Society of Anesthesiologists (ASA) III & IV.
* Local infection or sepsis at the site of injection.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  The degree of pain was assessed using the Visual analogue scale (VAS) [where (0 = no pain and 10 = severe pain)]. VAS was evaluated at 0, 2, 4, 6, 8, 12, 18, and 24 hours postoperatively.

SECONDARY OUTCOMES:
Duration of sensory block | Intraoperatively
  Duration of sensory block was assessed.
Time to first rescue analgesia | 48 hours postoperatively
  Time to first rescue analgesia was assessed from the end of surgery till first dose of pethidine administrated.
Total opioid consumption | 48 hours postoperatively
  If the Visual analogue scale (VAS) is ≥ 3, intravenous pethidine was given (0.5mg/kg).
Heart rate | 48 hours postoperatively
  Heart rate was recorded at baseline, after injection then every 30 min till the end of surgery and after surgery at 0, 2, 4, 6, 8, 12, 24 and 48 h.
Mean arterial pressure | 48 hours postoperatively
  Mean arterial pressure was recorded at baseline, after injection then every 30 min till the end of surgery and after surgery at 0, 2, 4, 6, 8, 12, 24 and 48 h.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.